CLINICAL TRIAL: NCT03602924
Title: Long-term Safety and Effectiveness in Motor and Non-motor Symptoms of Levodopa-carbidopa Intestinal Gel Infusion in Advanced Parkinson's Disease Patients With Motor Fluctuations
Brief Title: Long-term Safety and Effectiveness of Levodopa-carbidopa Intestinal Gel Infusion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)129/2008
Record Dates: First submitted 2018-06-27; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Parkinson Disease
Keywords: levodopa infusion
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Levodopa-carbidopa intestinal gel (LCIG) infusion has demonstrated to improve motor fluctuations. The aim of this study is to assess the long-term safety and effectiveness of LCIG infusion in advanced Parkinson's disease (PD) patients with motor fluctuations and its effect in non-motor symptoms.

DETAILED DESCRIPTION:
The following parameters were analyzed prior to LCIG treatment (at baseline), at months one, three, six and twelve, and every year afterwards over a 10-year period:

* Safety:

  - Adverse Events (AEs) related to percutaneous endoscopic gastrostomy (PEG) procedures and gastrostomy, infusion device, and treatment. Actions taken to solve them, and reasons for treatment discontinuation and withdrawal.
* Effectiveness:

  * Motor fluctuations: Off time in hours recorded in Parkinson's Disease Diary©.
  * Dyskinesia and other motor clinical aspects: evaluated with the Unified Parkinson's Disease Rating Scale (UPDRS) part IV, UPDRS part II in On and Off, UPDRS part III in On and Off, Hoehn and Yahr (H&Y) stage in On and Off and Schwab and England (S&E) scale.
  * Non-motor clinical aspects: cognitive function through Mini Mental State Examination (MMSE), and UPDRS part I, and relevant neuropsychiatric disorders.

The parameters analyzed in the three prospective substudies carried out in three subsets of this population, are described below:

Substudy 1 - Cognition and behavior assessment: Subgroup evaluated with a specific neuropsychological battery for assessment of cognition and behavior disorders prior to treatment (at baseline) and after 6 months of LCIG, by the same neuropsychologist at the same environmental conditions and in patients in phase On. The cognitive examination included: tests that assessed cognitive areas affected in PD according to the literature, psychometric tests with well-known parameters, tests that can be used in different types of populations (neurologic and psychiatric disorders, screening, etc.), tests suitable for a population with low educational and cultural level.

* Attentional function: Forward Digit Span test of Weschler Adult Intelligence Scale-Third Edition (WAIS III); Audio-verbal attentional capacity; and Stroop Color-Word test.
* Executive functions: Backward Digit Span of WAIS III; Audio-verbal working memory; Stroop-word and Stroop-color subtests; Response inhibition capacity; Controlled Oral Word-Association Test (FAS) of phonemic verbal fluency; Category Naming Test (Animals) of semantic verbal fluency.
* Visual-constructional visuospatial and visuoperceptual functions: Clock Drawing Test - (order and copy) -visual-constructional; Reading clocks - simple visuospatial ability; Luria test of overlapping figures - visual perceptive skills function.
* Memory and learning: Rey Auditory Verbal Learning Test (RAVLT) - Short and long term audio-verbal memory and recognition.
* Language: Boston Naming Test (BNT) - Title by visual comparison.
* Motor functions: Luria motor sequences - Voluntary motor control, Motor coordination.
* Mood: Beck depression inventory (BDI)
* Behavior: Neuropsychiatric Inventory (NPI) - Exploration of psychological and behavioral symptoms.

Substudy 2 - Quality of sleep: Subgroup evaluated with Epworth scale, fatigue scale, Pittsburg quality of sleep questionnaire, Beck Depression Inventory (BDI), and Hamilton anxiety scale, administered prior to treatment (at baseline) and 6 months after treatment. In addition, an overnight polysomnography (PSG) study was carried out at these timings.

Substudy 3 - Health status, QoL and caregiver burden: Subgroup evaluated for up to 12 months, with the Spanish version of the 39-items quality of life questionnaire in PD (PDQ-39, 0-156), health status questionnaires (EQ-5D, range 5-15; and EQ-VAS range 0-100), global clinical impression scale (CGI, range 1-7), and caregiver burden questionnaire or Zarit Burden index (ZBI, range 0-100). Assessments were done prior to treatment (at baseline), 1 week, 3 months, 6 months and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Parkinson's Desease (PD), diagnosed according to diagnostic criteria of the Brain Bank of London - United Kingdom Parkinson's disease Society Brain Bank (Gibb and Lees 1988; Hughes, Daniel et al. 1992; Calne, Snow et al 1992 ; Daniel i Lees 1993; Gelb, Oliver et al., 1999)
2. Patients with PD who respond to levodopa, according to the doctor's opinion. When the values of clinical scales with levodopa treatment achieve a 20-30% improvement in the scores of the Unified Parkinson's Disease Rating Scale (UPDRS). (UPDRS Off - UPDRS On) / UPDRS Off (Merello, Nouzeilles et al., 2002).
3. Patients with PD with a recognized Off and On status (motor fluctuations), confirmed by Parkinson's Disease Diary © (Hauser, Friedlander et al., 2000) at the start of the study (newspapers corresponding to 3 days preceding the initial visit).
4. Patients with PD in the advanced stage with severe motor fluctuations and dyskinesia induced by levodopa, poorly controlled with conventional optimized treatment.
5. Patients with PD in the advanced stage with severe motor fluctuations and dyskinesia induced by levodopa, poorly controlled with other complex treatments (such as apomorphine infusion pumps or ECP).
6. Patients with PD in the advanced state with serious motor fluctuations that present other non-motor complications such as depressive disorder, mild cognitive disorder, pulmonary control disorder, hallucinations and psychotic disorders and episodes of sleep, of moderate severity but , which excludes them from other alternatives to complex treatments, assisted with devices, second-line antiparkinsonians.
7. Patients who are capable, they or their responsible carers and assistants, to learn the treatment with levodopa intestinal infusion and the use of their devices and to guarantee their proper functioning and correct handling.
8. Patients with PD who have been indicated and who have agreed to begin treatment with levodopa intestinal infusion.
9. Patients who have included and granted their consent to participate in the prospective study of habitual clinical practice and have signed an informed consent form to participate in the study.
10. Women who have stopped menstruation naturally 24 months before, or are surgically sterile.
11. Women of childbearing age may participate in the study provided they use a contraceptive method acceptable from a medical point of view (a stable dose of contraceptive drug for at least 3 months or barrier methods: intrauterine device, diaphragm, or combination of condoms and spermicide).

    Women who are not nursing or are pregnant. Although no human teratogenicity has been described with levodopa treatment, and carbidopa does not cross the placental barrier and does not prevent these patients from interrupting oral levodopa during pregnancy (Merchant, Cohen et al., 1994; Ball i Sagar 1995; von Graevenitz, Shulman et al. 1996; Nomoto, Kaseda et al., 1997); In the event that it is considered GILC will start after pregnancy.
12. Patients attending the external consultation of the Neurology Service (Unit of Movement Disorders) at the Vall d'Hebron University Hospital.

Exclusion Criteria:

1. Patients who do not suffer from an idiopathic PD. That is, in which the diagnosis of PD is unclear or there is suspicion that there are other Parkinson's syndromes, such as secondary parkinsonism (caused by drugs, toxins, infectious agents, vascular disease, trauma or brain neoplasms), Parkinson plus syndromes (e.g., multi systemic atrophy, progressive supranuclear paralysis, corticosteroidal degeneration) or other neurodegenerative diseases.
2. Contraindications for the use of levodopa, such as narrow angle glaucoma, pheochromocytoma, Cushing syndrome or malignant melanoma history.
3. Treatment with non-selective MAO inhibitors and selective MAO type A inhibitors. These treatments should not be administered simultaneously with levodopa intestinal infusion. They must be taken down at least two weeks before the start of the treatment.
4. Psychiatric disorders, neurological or behavioral disorders that may interfere with the capacity of the subjects to give their informed consent to participate, or interfere with the performance or interpretation of the study; This category also includes serious hallucinations.
5. Cognitive deficiencies or dementias, defined as a score <24 in the Mini Mental State Exam (MMSE) (Folstein MF, Folstein et al., 1975) or that reach the criteria for the dementia of the Diagnostic and Statistical Manual of Fourth Mental Disorders (DSM-IV) (American Psychiatric Association 2000). Except for a compelling indication that the fluctuations are seriously impaired and correct and successful treatment and supervision can be guaranteed.
6. Abnormal laboratory data of clinical importance or any abnormal laboratory value that may interfere with the evaluation of safety according to the doctor.
7. Current indications of haematological, autoimmune, endocrine, cardiovascular, renal or gastrointestinal disorders of clinical importance that could interfere with the participation of the subject in the study.
8. Background or current suffering of gastrointestinal, liver, kidney or other pathology that may interfere with the absorption, distribution, metabolism or excretion of the study's drug or its evaluation, or interfere with the introduction of the probe system.
9. Medical, laboratory or surgical problems that the doctor considers to be of clinical importance.
10. Subjects in which the placement of a GEP-J probe is contraindicated for treatment with levodopa intestinal infusion or subjects considered to be of high risk for the GEP-J procedure, according to the evaluation performed by the gastroenterologist or the surgeon.

    The contraindications for the placement of the GEP-J probe include, among others, the following processes:
    1. Pathological changes in the gastric wall.
    2. Impossibility of joining the gastric wall and the abdominal wall.
    3. Blood clotting disorders: prothrombin activity less than 60% or INR of 1.4 and platelet count less than 80,000; Anticoagulant or antiaggregant treatment is not a contraindication but should be corrected and suspended before the procedure, due to the risk of bleeding.
    4. Pneumonia or severe respiratory failure. It has been suggested that a forced vital capacity of less than 1 liter and a pCO2 greater than 45 mmHg would be associated with an unacceptable mortality with the GEP procedure.
    5. Ascites
    6. Peritonitis
    7. Acute pancreatitis.
    8. Paralytic ileus.
    9. State of immunodeficiency, neutropenia, HIV, hypogammaglobulinemia, chronic steroid therapy.

    Except in cases where the indication of treatment with levodopa intestinal infusion is manifestly necessary and will be resorted to the implantation of a surgical gastrostomy.
11. Uncooperative attitude or reasonable probability that the subject does not comply with the treatment and the procedures of the study.
12. Subjects that do not provide their informed consent in writing to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with advanced PD, responders to levodopa and with disabling motor fluctuations. that fulfilled the UK Brain Bank criteria (Hughes et al., 1992) for the diagnosis of idiopathic PD and were experiencing severe motor fluctuations, which were debilitating in daily life, despite receiving optimized conventional oral medications. Patients had been previously treated with oral levodopa combined with entacapone, rasagiline, dopamine agonists and/or apomorphine injections. Patients with atypical parkinsonian features were not included.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-12-01 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in motor fluctuations of the Off time. | 10 years
  number of hours in Off time measured with Parkinson's Disease Diary © (Hauser, Friedlander et al., 2000). Changes will be compared to basal data.

SECONDARY OUTCOMES:
Change in proportion of the waking day with dyskinesia | 10 years
  Measured with the proportion of the day (in percentage) with dyskinesia. Responding to question 32 of Unified Parkinson's Disease Rating Scale (UPDRS) part IV categorizing 5 possible percentages: 0=0%, 1=1-25%, 2=26-50%, 3=51-75%, 4=76-100%. Understanding that the highest percentage indicates more time of the day in this period (historical information). Changes will be compared to basal data.
Change in severity of dyskinesia | 10 years
  Measured with the level of disability caused by dyskinesia. Responding to question 33 of the Unified Parkinson's Disease Rating Scale (UPDRS) part IV that categorizes in 0: they are not disabling, 1: mildly disabling, 2: moderately disabling, 3: severely disabling and 4: they produce total disability. Changes will be compared to basal data.
Change in parkinsonian motor symptoms assessed by the Unified Parkinson's Disease Rating Scale (UPDRS) | 10 years
  Measured with the Unified Parkinson's Disease Rating Scale (UPDRS) ranging from 0 (normal) to 199 (highest motor disability). Changes will be compared to basal data.
Change in Sleep Quality as assessed by Epworth Sleepines Scale (ESS) | 6 months
  Measured with Epworth Sleepines Scale (ESS) ranging from 0 (normal) to 24 (highest sleepiness). Changes will be compared to basal data.
Change in Sleep Quality as assessed by Pittsburgh Sleep Quality Index (PSQI) | 6 months
  Measured with Pittsburgh Sleep Quality Index (PSQI), ranging from 0 (healthier sleep quality) to 21 (worst sleep quality). Changes will be compared to basal data.
Total sleep time | One night at the sleep unit
  Total sleep time measured with an overnight polysomnography
Arousal index | One night at the sleep unit
  number of arousals/hour of sleep measured with an overnight polysomnography
Sleep architecture | One night at the sleep unit
  percentage of the different sleep phases measured with an overnight polysomnography
Change in cognitive function as assessed by the Unified Parkinson's Disease Rating Scale (UPDRS) | 6 months
  Measured with the Unified Parkinson's Disease Rating Scale (UPDRS) Part I (mentation, behavior and mood) ranging from 0 (normal) to 16 (highest cognitive function impaired). Changes will be compared to basal data.
Change in quality of life as assessed by 39-item Parkinson's disease Quality of Life Questionnaire Summary Index (PDQ-39) | 1 year
  Measured with of the 39-item Parkinson's disease Quality of Life Questionnaire Summary Index (PDQ-39) ranging from 0 (normal) to 100 (worst quality of life). Changes will be compared to basal data.
Change in caregiver burden as assessed by the Zarit caregiver Burden Index (ZBI) | 1 year
  Measured with of the Zarit caregiver Burden Index (ZBI) ranging from 0 (no overburden) to 110 (totally overburden). Changes will be compared to basal data.
Long term treatment safety as assessed by the ocurrence of serious advers events | 10 years
  Collecting adverse event that causes death, threatens life, requires hospitalization or prolongs hospitalization, causes disability or constitutes an important medical event.

CONTACTS AND LOCATIONS:
Overall Officials: Oriol de Fabregues, MD, PhD, Principal Investigator — neurologist
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Clinical Study report, results and statistical analysis, study protocol may be shared

REFERENCES:
- [Background] Antonini A, Isaias IU, Canesi M, Zibetti M, Mancini F, Manfredi L, Dal Fante M, Lopiano L, Pezzoli G. Duodenal levodopa infusion for advanced Parkinson's disease: 12-month treatment outcome. Mov Disord. 2007 Jun 15;22(8):1145-9. doi: 10.1002/mds.21500. PMID 17661426
- [Background] Antonini A, Yegin A, Preda C, Bergmann L, Poewe W; GLORIA study investigators and coordinators. Global long-term study on motor and non-motor symptoms and safety of levodopa-carbidopa intestinal gel in routine care of advanced Parkinson's disease patients; 12-month interim outcomes. Parkinsonism Relat Disord. 2015 Mar;21(3):231-5. doi: 10.1016/j.parkreldis.2014.12.012. Epub 2014 Dec 19. PMID 25585993
- [Background] Buongiorno M, Antonelli F, Camara A, Puente V, de Fabregues-Nebot O, Hernandez-Vara J, Calopa M, Pascual-Sedano B, Campolongo A, Valldeoriola F, Tolosa E, Kulisevsky J, Marti MJ. Long-term response to continuous duodenal infusion of levodopa/carbidopa gel in patients with advanced Parkinson disease: The Barcelona registry. Parkinsonism Relat Disord. 2015 Aug;21(8):871-6. doi: 10.1016/j.parkreldis.2015.05.014. Epub 2015 May 19. PMID 26003410
- [Background] Caceres-Redondo MT, Carrillo F, Lama MJ, Huertas-Fernandez I, Vargas-Gonzalez L, Carballo M, Mir P. Long-term levodopa/carbidopa intestinal gel in advanced Parkinson's disease. J Neurol. 2014 Mar;261(3):561-9. doi: 10.1007/s00415-013-7235-1. Epub 2014 Jan 30. PMID 24477490
- [Background] Catalan MJ, de Pablo-Fernandez E, Villanueva C, Fernandez-Diez S, Lapena-Montero T, Garcia-Ramos R, Lopez-Valdes E. Levodopa infusion improves impulsivity and dopamine dysregulation syndrome in Parkinson's disease. Mov Disord. 2013 Dec;28(14):2007-10. doi: 10.1002/mds.25636. Epub 2013 Oct 10. PMID 24123193
- [Background] Eggert K, Schrader C, Hahn M, Stamelou M, Russmann A, Dengler R, Oertel W, Odin P. Continuous jejunal levodopa infusion in patients with advanced parkinson disease: practical aspects and outcome of motor and non-motor complications. Clin Neuropharmacol. 2008 May-Jun;31(3):151-66. doi: 10.1097/wnf.0b013e31814b113e. PMID 18520982
- [Background] Fasano A, Ricciardi L, Lena F, Bentivoglio AR, Modugno N. Intrajejunal levodopa infusion in advanced Parkinson's disease: long-term effects on motor and non-motor symptoms and impact on patient's and caregiver's quality of life. Eur Rev Med Pharmacol Sci. 2012 Jan;16(1):79-89. PMID 22338551
- [Background] Fernandez HH, Standaert DG, Hauser RA, Lang AE, Fung VS, Klostermann F, Lew MF, Odin P, Steiger M, Yakupov EZ, Chouinard S, Suchowersky O, Dubow J, Hall CM, Chatamra K, Robieson WZ, Benesh JA, Espay AJ. Levodopa-carbidopa intestinal gel in advanced Parkinson's disease: final 12-month, open-label results. Mov Disord. 2015 Apr;30(4):500-9. doi: 10.1002/mds.26123. Epub 2014 Dec 24. PMID 25545465
- [Background] Nyholm D, Lewander T, Johansson A, Lewitt PA, Lundqvist C, Aquilonius SM. Enteral levodopa/carbidopa infusion in advanced Parkinson disease: long-term exposure. Clin Neuropharmacol. 2008 Mar-Apr;31(2):63-73. doi: 10.1097/WNF.0b013e3180ed449f. PMID 18382177
- [Background] Olanow CW, Kieburtz K, Odin P, Espay AJ, Standaert DG, Fernandez HH, Vanagunas A, Othman AA, Widnell KL, Robieson WZ, Pritchett Y, Chatamra K, Benesh J, Lenz RA, Antonini A; LCIG Horizon Study Group. Continuous intrajejunal infusion of levodopa-carbidopa intestinal gel for patients with advanced Parkinson's disease: a randomised, controlled, double-blind, double-dummy study. Lancet Neurol. 2014 Feb;13(2):141-9. doi: 10.1016/S1474-4422(13)70293-X. Epub 2013 Dec 20. PMID 24361112
- [Background] Puente V, De Fabregues O, Oliveras C, Ribera G, Pont-Sunyer C, Vivanco R, Cucurella G, Giralt E, Delgado T, Garcia C, Seoane A, Campo R. Eighteen month study of continuous intraduodenal levodopa infusion in patients with advanced Parkinson's disease: impact on control of fluctuations and quality of life. Parkinsonism Relat Disord. 2010 Mar;16(3):218-21. doi: 10.1016/j.parkreldis.2009.07.015. Epub 2009 Sep 16. PMID 19762271
- [Background] Zibetti M, Merola A, Artusi CA, Rizzi L, Angrisano S, Reggio D, De Angelis C, Rizzone M, Lopiano L. Levodopa/carbidopa intestinal gel infusion in advanced Parkinson's disease: a 7-year experience. Eur J Neurol. 2014 Feb;21(2):312-8. doi: 10.1111/ene.12309. Epub 2013 Dec 7. PMID 24313838